CLINICAL TRIAL: NCT04605471
Title: Safety Profile of Ultravist in Children and Elderly (UV Age)
Brief Title: A Study to Learn More About the Safety of Ultravist in Children and in the Elderly
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21494
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PMS I study: 'PMS I' was conducted in contrast-enhanced X-ray examination between June 1999 and November 2003 in 27 countries in Europe, Africa and Asia and comprised 74,717 patients of which 2,172 were children and 32,103 were elderly patients.
  Ref. Kopp AF, Mortele KJ, Cho YD, Palkowitsch P, Bettmann MA, Claussen CD. Prevalence of acute reactions to iopromide: postmarketing surveillance study of 74,717 patients. Acta Radiol. 2008;49(8):902-11.
  Interventions: Drug: Iopromide(Ultravist, BAY86-4877)
- IMAGE study: 'IMAGE' consists of 44,835 patients with contrast-enhanced X-ray examination and was conducted in 21 European and Asian countries from February 2008 to September 2009, 1,451 patients were children, and 15,654 were elderly patients.
  Ref. Palkowitsch P, Lengsfeld P, Stauch K, Heinsohn C, Kwon ST, Zhang SX, et al. Safety and diagnostic image quality of iopromide: results of a large non-interventional observational study of European and Asian patients (IMAGE). Acta Radiol. 2012;53(2):179-86.
  Interventions: Drug: Iopromide(Ultravist, BAY86-4877)
- TRUST study: 'TRUST' assessed the safety and tolerability of Ultravist in patients undergoing cardiac catheterization. It was conducted from August 2010 to September 2011 in China and included 17,513 patients of which 12 were children and 8,918 were elderly patients.
  Ref. Chen JY, Liu Y, Zhou YL, Tan N, Zhang B, Chen PY, et al. Safety and tolerability of iopromide in patients undergoing cardiac catheterization: real-world multicenter experience with 17,513 patients from the TRUST trial. Int J Cardiovasc Imaging. 2015;31(7):1281-91.
  Interventions: Drug: Iopromide(Ultravist, BAY86-4877)
- Ultravist in CT study: 'Ultravist in CT' was performed with focus on contrast-enhanced CT examination between November 2006 and December 2008 and included 15,168 patients in Germany, Iran, Romania and Saudi Arabia. A total of 417 patients were children, 7,453 were elderly patients.
  Ref. Palkowitsch PK, Bostelmann S, Lengsfeld P. Safety and tolerability of iopromide intravascular use: a pooled analysis of three non-interventional studies in 132,012 patients. Acta Radiol. 2014;55(6):707-14.
  Interventions: Drug: Iopromide(Ultravist, BAY86-4877)

INTERVENTIONS:
Drug: Iopromide(Ultravist, BAY86-4877) — The study will be conducted by using pooled data of four company sponsored non-interventional studies with iopromide.

SUMMARY:
Ultravist is an iodine-based contrast agent that helps to make medical imaging scans clearer. It is also called iopromide, and it is available for doctors to give patients before they have scans. Even after a treatment or substance has been approved for use, researchers continue to study it to learn more about its safety.

Researchers have done studies on the safety of Ultravist, but they want to learn more about specific medical problems called hypersensitivity reactions (HSRs). These are undesirable immune system reactions to the study drug. In this study, the researchers will compare the risk of HSRs in children and in the elderly to the risk of HSRs in middle aged adults.

The researchers will look at information about medical problems that happened in people in 4 other studies. These studies are called PMS I, IMAGE, TRUST, and Ultravist in CT. A total of about 139,000 people will be included in this study.

All of the people in the earlier 4 studies received Ultravist as an injection into the vein or artery before having a scan. In this study, the researchers will compare the number of children, middle aged adults, and elderly patients who had HSRs after receiving Ultravist.

ELIGIBILITY:
Inclusion Criteria:

* We included patients of all age groups which were referred to a iodine-based contrast-enhanced procedure of any body part.

Exclusion Criteria:

* Patients with missing age, sex or who did not receive Ultravist 300 or 370 were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients who received a contrast enhanced X-ray based examination with Ultravist for various clinical reasons
Sampling Method: Non-Probability Sample
Enrollment: 132850 (Actual)
Dates: Start 2020-10-31 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with hypersensitivity reactions to Ultravist in children and elderly patients compared to middle-age adults | Analysis will be done in 2 months

SECONDARY OUTCOMES:
Profile of HSRs (hypersensitivity reactions) in the three age groups | Analysis will be done in 2 months
General reported ADR (adverse drug reactions) profile in the three age groups | Analysis will be done in 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Four company sponsored non-interventional studies with iopromide, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Endrikat J, Chernova J, Gerlinger C, Pracz M, Lengsfeld P, Bhatti A, Michel A. Risk of Hypersensitivity Reactions to Iopromide in Children and Elderly: An Analysis of 132,850 Patients From 4 Observational Studies and Pharmacovigilance Covering >288 Million Administrations. Invest Radiol. 2022 May 1;57(5):318-326. doi: 10.1097/RLI.0000000000000840. PMID 34860739